CLINICAL TRIAL: NCT02371395
Title: Validation of RealAmp Method for the Diagnosis of Malaria in Endemic Areas of Brazil
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Evandro Chagas Institute of Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: 6619
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2015-05

CONDITIONS: Malaria Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Realtime amplification (RealAmp) — Molecular assay for the diagnosis of malaria.

SUMMARY:
Worldwide, approximately 2 billion people live in areas at risk for malaria with morbidity surpassing 250 million cases, with approximately 800,000 deaths, per year. Of the four species of malaria parasites that cause human infection, P. falciparum is responsible for the majority of severe malaria cases followed by P. vivax. Early and accurate diagnosis is essential for prompt and correct treatment, which can reduce the death rate and interrupt transmission. Currently, conventional methods for the diagnosis of malaria include microscopic examination of thin and thick blood smears and rapid diagnostic tests (RDTs). Light microscopy in practice typically detects parasitemia as low as 100 parasites/µl and it can differentiate species. The advantage of microscopy includes the ability to estimate parasitemia, the possibility to identify parasite stages, including gametocytes, and its low cost. However, this method is labor intensive, difficult to standardize, and requires well-trained microscopists. The majority of RDTs are based on detection of P. falciparum histidine-rich protein 2 (HRP-2) antigen and do not detect all malaria species. RDTs that detect lactose dehydrogenase (LDH) and aldolase generally broadly react with all four species of malaria parasites and therefore cannot differentiate among the species although efforts are underway to improve their performance for species detection. In settings where multiple malaria species co-circulate, molecular methods may be more reliable than microscopy and RDTs in accurately diagnosing the species of malaria parasites with low parasitemias. However, conventional molecular methods, such as nested polymerase chain reaction (nested PCR) or real-time PCR, are technically challenging and resource intensive and are generally restricted to reference laboratories due to the need for well-equipped laboratories. Recently, new molecular methods that can be used in field settings have been developed and this opens up new opportunities for exploring molecular tools for malaria diagnosis in endemic countries. With the objective of facilitating use of molecular tools for malaria control programs, the malaria laboratory at the Centers for Disease Control and Prevention (CDC) in Atlanta, USA developed a simple isothermal molecular method called Real-Time Fluorescence Loop-Mediated Isothermal Amplification (RealAmp) for the diagnosis of malaria. Currently, RealAmp primers exist for detecting the Plasmodium genus and the detection of P. falciparum and P. vivax species. The RealAmp method has great potential as a molecular tool for the diagnosis of malaria in the field (and other infections of major public health impact, such as HIV and tuberculosis). It can provide an alternative to conventional PCR-based diagnostic methods for field use in clinical and operational programs. The objective of this proposal is to validate the sensitivity of RealAmp for detection of malaria parasites in blood spots from patients with clinical diagnosis of malaria in two endemic states of Brazil with co-circulation of P. falciparum and P. vivax. In this evaluation, RealAmp and microscopic examination will be compared to a real-time PCR method as a reference test.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years
* Signed informed consent for patients 18 years and older
* Signed parental/guardian consent form and assent from the patient (for those less than 18 years)
* Documented fever (auxiliary temperature greater than 37.5C) or self-reported fever in previous 24 hours in the absence of another obvious cause of fever
* First visit for current illness at the diagnostic post

Exclusion Criteria:

* Absence of fever or no history of fever
* Follow-up visit for the current illness
* No consent/assent to participate
* Antimalarial treatment use in previous 30 days

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with fever who present for malaria diagnosis and regular health posts.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Macedo de Oliveira, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Hospital do Jurua, Cruzeiro do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Suspected Malaria (Fever): This was a study of enrolling patients with fever or history of fever for malaria testing. A total of 1,000 samples were collected from patients in Cruzeiro do Sul, Acre state from January to June, 2015.
Period: Overall Study
Arm/Group | Patients With Suspected Malaria (Fever)
Started | 1000
Completed | 1000
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: This was a study of enrolling patients with fever or history of fever for malaria testing. A total of 1,000 samples were collected from patients in Cruzeiro do Sul, Acre state from January to June, 2015.
Arm/Group | Single Arm
Number analyzed (Participants) | 1000
Age, Continuous [Median (Full Range); unit: years] | 29.5 [7 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 551
  Male | 449
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 1000

OUTCOME MEASURES:

1. Primary Outcome: Malaria Diagnosis Using RealAmp and Microscopy.
Description: These are the results of the different tests used in the evaluation.
Time Frame: 12 months
Population: Those were patients presenting with suspected malaria.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 1000
Participants
  Number of positive samples by local microscopy: P. falciparum | 42
  Number of positive samples by local microscopy: P. vivax | 153
  Number of positive samples by local microscopy: Mixed infection | 0
  Number of positive samples by local microscopy: Species unidentified | 1
  Number of positive samples by local microscopy: Negative | 804
  Number of positive samples by study microscopy: P. falciparum | 56
  Number of positive samples by study microscopy: P. vivax | 169
  Number of positive samples by study microscopy: Mixed infection | 1
  Number of positive samples by study microscopy: Species unidentified | 0
  Number of positive samples by study microscopy: Negative | 774
  Number of positive samples by RealAmp: P. falciparum | 55
  Number of positive samples by RealAmp: P. vivax | 181
  Number of positive samples by RealAmp: Mixed infection | 0
  Number of positive samples by RealAmp: Species unidentified | 3
  Number of positive samples by RealAmp: Negative | 761
  Number of positive samples by reference test: P. falciparum | 48
  Number of positive samples by reference test: P. vivax | 152
  Number of positive samples by reference test: Mixed infection | 20
  Number of positive samples by reference test: Species unidentified | 0
  Number of positive samples by reference test: Negative | 780

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/1000
Other Adverse Events (participants affected / at risk) | 0/1000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No